CLINICAL TRIAL: NCT00669305
Title: Bone Marrow for Hemoglobinopathy Research
Status: Completed | Type: Observational
Sponsor: St. Jude Children's Research Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Assisi Foundation (Other); University of Tennessee (Other)
Responsible Party: Sponsor
Other Study IDs: BMR; U54HL070590 (NIH); P01HL053749 (NIH); 201003 (Other: Doris Duke Foundation)
Record Dates: First submitted 2008-04-28; First posted 2008-04-30 (Estimated); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Sickle Cell Anemia; Thalassemia
Keywords: Genetics; Blood cells; Vector-mediated gene transfer; Bone marrow; CD34 cells
MeSH Terms: conditions — Anemia, Sickle Cell; Thalassemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Stem Cells through Bone Marrow Aspiration
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort 1: Human participants affected with sickle cell disease or thalassemia will donate bone marrow for use in experimental models

SUMMARY:
Human participants affected with sickle cell disease or thalassemia will donate bone marrow for use in experimental laboratory models to study potential new treatments. This is an observational study using bone marrow from human participants. The investigators will use sickle cell and thalassemia mouse models to observe and evaluate the possibility of correcting these disorders through genetic alterations or drug treatment.

DETAILED DESCRIPTION:
These studies are designed to evaluate the potential of retroviral vector mediated gene transfer, gene editing, or drug treatment to correct the pathophysiology of sickle cell anemia and β-thalassemia. CD34+ cells purified from bone marrow of research participants with a sickle cell syndrome or a thalassemia syndrome will be subjected to genetic editing, drug treatment, or transduced with retroviral vectors containing γ-globin coding sequences under the control of the β-globin gene promoter and including various regulatory elements chosen to enhance gene expression and to insulate regulatory elements from cellular genes at or near the integration sites. The efficiency of gene transfer and the function of the globin transgene will be evaluated in erythroid cells derived from transduced progenitors and from the progenitors in the bone marrow of immunodeficient mice engrafted with transduced, primitive hematopoietic cells. The hypothesis to be tested in this research is that a gene therapy vector, gene editing strategy, or drug modality can be designed to achieve a potentially therapeutic level of globin gene expression in maturing erythroid cells.

ELIGIBILITY:
Inclusion Criteria:

* Patients with homozygous S/S disease or doubly heterozygous for S and β thalassemia who are 2 years or older are eligible. Patients with HbE- β- thalassemia or homozygous (severe) β-thalassemia are also eligible. Patients with thalassemia include those who are transfusion dependent (major) or severely anemic but relatively transfusion independent (intermedia). Diagnostic criteria include standard hematological parameters, red cell indices, hemoglobin electrophoresis and quantitative determination of HbF and HbA2.
* Patients are eligible for participation in the protocol only if they are currently clinically stable and have been free of all acute disease manifestations for a minimum of 14 days.
* Patients may participate while continuing their current therapeutic regimen including regular transfusion therapy or hydroxyurea administration.
* In general, two categories of patients will be considered as research participants in this protocol.

  1. Patients who are 18 years or older and therefore able to provide informed consent will be eligible. Such individuals will be recruited from among patients followed at SJCRH. In addition, individuals followed in an outside clinic who are recruited will be asked to come to the Hematology Clinic at SJCRH to enroll and have the procedure performed. Alternatively, if a patient who is 18 or older is to undergo a diagnostic or surgical procedure under general anesthesia, and they agree to participate in the study, the bone marrow aspirate will be obtained at that time.
  2. Patients between the ages of 2 and 17 years who are scheduled for a diagnostic or surgical procedure at SJCRH or LeBonheur Children's Medical Center for which sedation or general anesthesia is indicated will be eligible for protocol enrollment. A bone marrow aspiration will be performed during the sedation or general anesthesia for the diagnostic or surgical procedure.

Exclusion Criteria:

* Active, acute manifestations of sickle cell disease including painful crisis, acute chest syndrome, cerebrovascular events or active infection.
* Pregnant women will not be eligible for study enrollment.
* Inability or unwillingness of the research participant or legal guardian/representative to give written informed consent will preclude enrollment on this research protocol.
* Platelet count < 150,000/mm^3
* Neutrophil count < 2000/mm^3 (unless on hydroxyurea therapy)
* Neutrophil count < 1000/mm^3 for patients on hydroxyurea therapy
* Prothrombin Time > 17 seconds
* Partial thromboplastin Time > 43 seconds
* History of excessive bleeding in the context of previous procedures including surgery and dental extractions

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Sickle Cell Anemia or Thalassemia
Sampling Method: Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2008-05-15 (Actual); Primary Completion 2019-08-29 (Actual); Study Completion 2019-08-29 (Actual)

PRIMARY OUTCOMES:
Percentage of successful achievement of therapeutic level in mouse models resulting from retroviral vector mediated gene transfer, gene editing or drug treatment. | 4 years
  The specific hypothesis to be tested is that a gene therapy vector, gene editing strategy, or drug modality can be designed that achieves a therapeutic level of globin production in transduced cells in mouse models.

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell J. Weiss, MD, PhD, Principal Investigator — St. Jude Children's Research Hospital
Locations (1):
- St. Jude Children's Research Hospital, Memphis, Tennessee, United States

REFERENCES:
- See also: St. Jude Children's Research Hospital — http://www.stjude.org
- See also: Clinical Trials Open at St. Jude — http://www.stjude.org/protocols